CLINICAL TRIAL: NCT04596722
Title: Prospective Randomized Double-Blind Placebo Controlled Study of Oral Pomella on the Microbiome and Skin Biophysical Properties
Brief Title: Oral Pomegranate Extract on the Microbiome and Skin Biophysical Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Verdure Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POM01
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Human Microbiome
Keywords: gut microbiome; polyphenols; skin; dermatology; pomegranate extract; punicalagins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned Interventions (Active Comparator): oral active pomella taken by mouth once per day
  Interventions: Dietary Supplement: Pomella
- Placebo (Placebo Comparator): oral placebo taken by mouth once per day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Pomella — Pomella® Pomegranate Whole Fruit Extract containing 75 mg punicalagin in white/white HPMC size "1" capsules packed in white color HDPE bottle of 30 counts
  Arms: Assigned Interventions
Other: Placebo — White/white HPMC size "1" capsules each containing 97.67% Maltodextrin, 0.10% Tartrazine color, 0.22% Brown Color, 2.01% Aerosil packed in white color HDPE bottle of 30 counts
  Arms: Placebo

SUMMARY:
Pomegranate extract (Pomella) is well known for its antioxidant properties due to its phenolic compounds. It has also been shown to increase the amount of short chain fatty acid producing Lactobacillus and Bifidobacteria genera. Short chain fatty acids are thought to have an anti-inflammatory effect on the sebaceous glands. Previous studies have concluded that pomegranate extract may act as a prebiotic in the body and subsequently increasing the gastrointestinal microbial diversity and by producing short chain fatty acids that may have systemic beneficial effects especially on the skin.

Therefore, the aim of this study is to assess how Pomella alters the gut microbiome and the blood level of short chain fatty acids in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 25-55
2. Must be willing to comply with all protocol requirements
3. Must be willing to have flash photo facial images taken with the imaging systems
4. Males must be willing to shave any facial hair

Exclusion Criteria:

1. Any systemic or antibiotics (injected or oral) within 6 months of starting study
2. Any topical antibiotic or benzoyl peroxide within 1 month of starting study or any subject unwilling to refrain from washout of topical antibacterial or benzoyl peroxide ingredient.
3. No intake of alcohol or tea throughout the duration of the study.
4. No more than 1 8 oz cup of coffee per week throughout the duration of the study.
5. No more than 1 cup of berries (strawberries, blueberries, raspberries, blackberries, etc.) per week throughout the duration of the study.
6. No intake of pomegranate, or pomegranate-containing drinks throughout the duration of the study.
7. No intake of chocolate (in any form) throughout the duration of the study.
8. No more than 1 cup of fermented dairy products per week throughout the duration of the study.
9. Any oral probiotic or prebiotic supplementation within past 1 month
10. Subjects must have no history of malignancy or cancer or diagnosis of gastrointestinal inflammatory diseases, no history or diagnosis of epilepsy, no history or diagnosis of immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus, rheumatoid arthritis)
11. Has a condition or is on medication the investigator and/or designee believe could jeopardize the safety of the subject, interfere with the evaluation, or confound the interpretation of the study results
12. Women who have been pregnant in the last three months, are pregnant, preparing to be pregnant or lactating.
13. Is participating in a concurrent clinical research study or has participated in an acne or other facial study at this or any other facility in the past 4 weeks
14. Those with BMI higher than 35 kg/m²
15. Commencement of a new diet (such as the ketogenic diet) or supplements within the 1 month prior to initiating participation, at the discretion of the investigator.
16. Use of medications that alter blood lipids, such as statins and anti-hyperlipidemic medications
17. Is participating in or has participated in a facial study at this or any other facility in the past 4 weeks. Participation in survey-based studies are approved at the discretion of the investigator.
18. Has a skin disease on face that will interfere with image collection and assessment in the opinion of the investigator
19. Refusal to shave or remove facial hair that may interfere with image collection and assessment.
20. Persons unwilling to avoid the following during the 4 weeks prior and during the duration of the study: self-tanning, spa tanning, sun tanning, or artificial tanning.
21. Planned vacation to sunny destination with the intention of sun tanning during the duration of the study.
22. Persons who regularly undergo sauna treatments (dry or wet) or who swim daily.
23. Known allergy or irritation to the supplement or facial products utilized in the study
24. Current tobacco smokers, OR those that have smoked tobacco over the past year, OR a 5 year-pack year history of smoking tobacco
25. Prisoners
26. Adults unable to consent
27. Vegans

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Shift in Gut Microbiome Diversity | 4 weeks
  Stool is collected and analyzed for species of bacteria through nucleic acid sequencing.

SECONDARY OUTCOMES:
Gut Microbiome Changes- Abundance and Presence of Short Chain Fatty Acid producing Bacteria | 4 weeks
  Stool is collected and analyzed for species of bacteria through nucleic acid sequencing.
Safety Assessment for GI Distress | 4 weeks
  Subjective GI based Questionnaire that will assess for distress (one combined metric that accounts for stooling, gas, and discomfort)
Change in Skin Brightness - Device based | 4 weeks
  SkinColorCatch colorimeter RGB range: 25-246 per channel
Change in Sebum Excretion Rate | 4 weeks
  Delfin Sebumeter: 0-150 micrograms/cm^2
Change in Transepidermal Water Loss | 4 weeks
  Delfin Vapometer 0-300g/m^2h; Delfin MoisturemeterSC 0-150
Change in the Appearance of Facial Redness and Facial Skin Tone | 4 weeks
  SkinColorCatch colorimeter RGB range: 25-246 per channel; BTBP Clarity Mini 3D_V5 camera
Shift in the Blood Short Chain Fatty Acid Levels | 4 weeks
  Short chain fatty acids are measured from a venipuncture
Change in skin brightness - image based | 4 weeks
  BTBP Clarity Mini 3D Camera

OTHER OUTCOMES:
Change in Skin Microbiome Diversity | 4 weeks
  The alpha and beta diversity of facial skin microbiome collections will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States